CLINICAL TRIAL: NCT00910793
Title: Open-Label, Prospective Study to Assess the Effects of Formoterol and Beclometasone Dipropionate Combination Therapy on Central and Peripheral Airway Dimensions in Asthmatic Patients
Brief Title: Study to Assess the Effect of Formoterol and Beclomethasone Dipropionate in Asthmatic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wilfried De Backer (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Wilfried De Backer, MD PhD, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PML_DOC_0802; Eudract number: 2008-002391-97
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Beclomethasone Dipropionate; Computational Fluid Dynamics; Functional Imaging; Central and Peripheral Airways
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inuvair (Other)
  Interventions: Drug: Inuvair

INTERVENTIONS:
Drug: Inuvair — 6 µg formoterol and 100 µg beclometasone dipropionate combination spray pMDI aerosol

SUMMARY:
The objective of this study is to evaluate the effect of the combination of formoterol and beclometasone dipropionate on central and peripheral airway dimensions in asthmatic patients using Computational Fluid Dynamics (CFD). Further more, the effect of this combination therapy on exhaled NO, lung function (spirometry, body plethysmography, diffusion and resistance) and subjective asthma control score as well as the safety of this combination will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asthma as defined by the current Global INitiative for Asthma (GINA) guidelines:
* Male or female patients aged ≥18 years
* Patients with a documented positive response to the reversibility test within the 12 months preceding the screening visit or performed at screening visit after a wash-out of 2 days for long acting β2 agonists or a documented positive response to the methacholine challenge test
* Patients with a co-operative attitude and ability to be trained to correctly use the pressurized Metered Dose Inhaler (pMDI)
* Written informed consent obtained

Exclusion Criteria:

* Pregnant or lactating females or females at risk of pregnancy
* Inability to carry out pulmonary function testing
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) as defined by the current Global initiative for chronic Obstructive Lung Disease (GOLD) guidelines
* History of near fatal asthma
* Hospitalization due to asthma or symptomatic infection of the airways in the previous 8 weeks
* Current smokers or recent (less than one year) ex-smokers, defined as smoking at least 10 cigarettes/day
* Patients with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study
* Patients with a QTc interval (Bazett's formula) at the screening visit Electrocardiogram (ECG) test >450 msec
* Cancer or any other chronic disease with poor prognosis and /or affecting patient status
* History of alcohol or drug abuse
* Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients
* Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
* Patients who received any investigational new drug within the last 8 weeks prior to the screening visit
* Patients treated with any non-permitted concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Differences in airway dimension | airway dimension will be measured at visit 2 and visit 7
  The primary objective of this study is to evaluate the effect of the combination therapy on central and peripheral airway dimensions with CFD. The following primary outcome parameters will be determined:
  * Total airway resistance for the segmented airways
  * Peripheral airway resistance(from 4th bifurcation on) for the segmented airways
  * Total airway volume for the segmented airways
  * Peripheral airway volume (from the 4th bifurcation on) for the segmented airways
  * Relative compliance for each lobe
  * Density of the lung parenchyma given per predefined lung zone

SECONDARY OUTCOMES:
Lung function tests: dynamic lung volumes, static lung volumes and airway resistances | lung function tests will be perfomed at te following visits: screening, visit 1 (2 weeks after screening), visit 3 (6 weeks after screening), visit 5 (14 weeks after screening) and visit 7 (26 weeks after screening)
  The secondary outcome parameters that will be obtained with the lung function tests are:
  * Dynamic lung volumes: Forced Expiratory Volume in 1 sec (FEV1), Forced Vital Capacity (FVC), Peak Expiratory Flow (PEF),Maximum expiratory flow when 50% of the FVC remain to be exhaled (MEF50) , Maximum expiratory flow when 25% of the FVC remain to be exhaled (MEF25)
  * Static lung volumes: Vital Capacity (VC),Inspiratory Vital Capacity (IVC), Functional Residual Capacity (FCR), Total Lung Capacity (TLC)
  * Airway resistances: Airway Resistance (Raw), Specific Airway Conductance(SGaw) (based on body plethysmography)
Subjective asthma control score | Asthma Control Test (ACT) will be performed on visit 1, 2, 3, 5 and 7
  Asthma control scores will be obtained with the Dutch Asthma Control Test.
Exhaled Nitric Oxide (NO) | Exhaled NO will be measured on visit 2, 3, 5 and 7
Adverse events as a measure of safety | Follow up of adverse events will be done during the entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Antwerp, Belgium